CLINICAL TRIAL: NCT00097240
Title: The Raptiva Pregnancy Registry: An Observational Study of the Use and Safety of Raptiva (Efalizumab) During Pregnancy
Brief Title: An Observational Study of the Use and Safety of Raptiva During Pregnancy (FOLLOW)
Acronym: FOLLOW
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Other Study IDs: ACD3100g
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Psoriasis; Pregnancy
Keywords: FOLLOW; Psoriasis; Pregnancy
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Raptiva Pregnancy Registry was a prospective observational study established to obtain data on pregnancy outcomes of women who were exposed to Raptiva.

ELIGIBILITY:
Any patient who has used Raptiva within 6 weeks prior to conception or during her pregnancy may be included in the Registry. Enrollment is based on Raptiva exposure, whether inadvertent or deliberate, in relation to pregnancy. Enrollment should occur as early as possible during the pregnancy and must occur prior to knowledge of pregnancy outcome.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women solicited through advertising, physician and patient awareness, and other programs.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2005-01; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D, Study Director — Genentech, Inc.
Locations (1):
- FOLLOW Raptiva Pregnancy Registry, Morrisville, North Carolina, United States